CLINICAL TRIAL: NCT04637607
Title: Immediate Effect of Non-invasive Auricular Acupoint Stimulation on the Performance and Meridian Activities of Archery Athletes- a Protocol for Randomized Controlled Trial
Brief Title: Immediate Effect of Non-invasive Auricular Acupoint Stimulation for the Performance and the Meridian Activities of Archery Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CMRPG8J0941
Record Dates: First submitted 2020-11-04; First posted 2020-11-20 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2020-11

CONDITIONS: Stress, Physiological; Sport Injury
Keywords: archery; Ryodoraku; heart rate variability; auricular acupoint

STUDY DESIGN:
Intervention Model Description: The study recruited the archery players in school teams among junior high, senior high schools, and colleges.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants were randomly assigned to the treatment group and the control group. The Ear-Acupressure group received the seeds attached by 3M tap to the auricular acupoints. The Sham-Acupressure group received sham acupoint stimulation, on the same points, but only with 3M tap. The procedure was then switched to perform cross-over study design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ear-Acupressure Group (Experimental): The subjects will receive true auricular acupoints stimulation with the attachment of Vaccaria seeds during the first round of play. After finishing the first round, the subjects will receive sham auricular acupoints stimulation.
  Interventions: Other: Auricular acupoints stimulation
- Sham-Acupressure Group (Sham Comparator): The subjects will receive sham auricular acupoints stimulation with the attachment of Vaccaria seeds during the first round of play. After finishing the first round, the subjects will receive true auricular acupoints stimulation. (Crossover)
  Interventions: Other: Auricular acupoints stimulation

INTERVENTIONS:
Other: Auricular acupoints stimulation — Noninvasive auricular acupoints stimulation with seeds

SUMMARY:
In our hypothesis, auricular acupoint stimulation might improve the attention and heart rate variability in archery athletes. The meridian activities regarding the attention and action in Chinese medicine systems might be influenced.

DETAILED DESCRIPTION:
During the execution of archery, attention is the key of performance in elite players, especially in the initial period.

Auricular acupoint stimulation is one of the therapeutic methods of traditional Chinese medicine. It is widely applied in various diseases. Researches had concluded the use of auricular acupoint stimulation on amplifying the anesthesia effect, weight reduction and the cessation of substance abuse. This study aimed to investigate the immediate effect of non-invasive auricular acupoint stimulation on the performance and the meridian activities of archery athletes.

The investigators will collect the meridian activities and balance index with Ryodoraku device, the continuous heart rate record and the scores of the two sections as the performance. The participants will rate their attention and fatigue levels through filling the self-reported questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Health volunteers, age between 13-26 years old
* Received training of archery for more than one year

Exclusion Criteria:

* History of psychiatric disorders
* History of cardiovascular diseases
* Previous operation history of dominant hand
* Unwilling or unable to sign the informed consent of this study

Ages: 13 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
The change of meridian activities | Baseline, one hour, two hours
  The meridian activities and balance index were measured and calculated with Ryodoraku device. (Meridian Energy Analysis Device, MEAD, medpex, Taiwan) The activity will be shown by numbers which were calculated by the skin electric resistance. The higher the number is, the higher meridian activity is presented.
The change of heart rate variability | Two and half hours, keep recording during the whole process
  Analyzed by continuous heart rate recording with heart rate monitor (Garmin, the U.S.)
The change of Checklist Individual Strength, CIS | Baseline, one hour, two hours
  The self-reported attention and fatigue questionnaire which is composed with 30 items. Each item ranks from zero to five. Higher scores indicated higher distraction and fatigue levels.
The change of Visual Display Terminals visual syndrome, VDTs fatigue scale | Baseline, one hour, two hours
  The self-reported attention and fatigue questionnaire which focus at visual syndrome. VDTs fatigue scale is been applied and standarized by Japanese Ministry of Health, Labor and Welfare survey results, 2004. VDTs fatigue scale is composed with 13 items. Each item ranks from zero to five. Higher scores indicated higher distraction and fatigue levels.

SECONDARY OUTCOMES:
The change of motion stabilization | Two and half hours, keep recording during the whole process
  Recorded and analyzed by the WIMU PRO (RealTrack Systems, Almería, Spain) The bluetooth data will be collected and analyzed to show the motion characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: CHUN EN KUO, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Department of Chinese Medicine, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hatfield BD, Landers DM, Ray WJ. Cardiovascular-CNS interactions during a self-paced, intentional attentive state: elite marksmanship performance. Psychophysiology. 1987 Sep;24(5):542-9. doi: 10.1111/j.1469-8986.1987.tb00335.x. No abstract available. PMID 3685234
- [Result] Carrillo AE, Christodoulou VX, Koutedakis Y, Flouris AD. Autonomic nervous system modulation during an archery competition in novice and experienced adolescent archers. J Sports Sci. 2011 Jun;29(9):913-7. doi: 10.1080/02640414.2011.568514. PMID 21547837
- [Derived] Tsai YH, Wu SY, Hu WL, Lai YR, Tsao Y, Yen KT, Lin CH, Kuo CA. Immediate effect of non-invasive auricular acupoint stimulation on the performance and meridian activities of archery athletes: A protocol for randomized controlled trial. Medicine (Baltimore). 2021 Feb 26;100(8):e24753. doi: 10.1097/MD.0000000000024753. PMID 33663090